CLINICAL TRIAL: NCT01668433
Title: Open Label Randomized Controlled Trial Pharmacokinetic and Vitro Transmission Blocking Activities Study of Primaquine Compare to Methylene Blue in Healthy Volunteer Both G6PD Normal and G6PD Deficiency
Brief Title: Pharmacokinetic and in Vitro Transmission Blocking Activities Study of Primaquine Compare to Methylene Blue in Healthy Volunteer Both G6PD Normal and G6PD Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FTM1201
Record Dates: First submitted 2012-08-01; First posted 2012-08-20 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: G6PD Normal; G6PD Deficient; Healthy
Keywords: G6PD; Primaquine; Methylene blue
MeSH Terms: interventions — Clinical Protocols; Primaquine; Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G6PD Normal (Active Comparator): Subjects will be given either primaquine, 45 mg single dose or methylene blue, 600 mg single dose with a washout period of 7 days then followed by either methylene blue, 600 mg single dose or primaquine, 45 mg single dose.
  Interventions: Drug: Regimens (Primaquine, Methylene blue)
- G6PD deficiency (Experimental): Subjects will be given either primaquine, 45 mg single dose or methylene blue, 600 mg single dose with a washout period of 7 days then followed by either methylene blue, 600 mg single dose or primaquine, 45 mg single dose.
  Interventions: Drug: Regimens (Primaquine, Methylene blue)

INTERVENTIONS:
Drug: Regimens (Primaquine, Methylene blue) — Primaquine 45 mg single dose Or Methylene Blue 600 mg single dose followed by Methylene Blue 600 mg single dose or Primaquine 45 mg single dose.

SUMMARY:
The emergence of partial artemisinin resistance in Plasmodium falciparum on the Cambodia-Thai border and more recently on the Myanmar-Thai border jeopardizes the renewed global efforts of control and elimination of malaria. Containment of this severe threat requires reduction of transmission of the resistant phenotype by adding gametocytocidal drugs to the treatment of falciparum malaria. Mathematical models also predict that transmission blocking will be required if the goal of malaria elimination is to be achieved. The only drug currently available with strong gametocytocidal properties against the more mature gametocytes is primaquine. However, the oxidative properties of primaquine readily causes acute haemolysis in glucose 6 phosphate dehydrogenase (G6PD) deficiency, the degree of which appears to be inversely related to G6PD enzyme activity. Because of these safety concerns, primaquine is not widely deployed in treatment regimens for falciparum malaria, even in areas with documented artemisinin resistance. Methylene blue, which does not exert its action through an oxidative mechanism, is a promising alternative as a gametocytocidal adjuvant to artemisinin combination therapies (ACTs). Paul Ehrlich discovered methylene blue as the first synthetic drug ever to treat malaria. In contrast with primaquine, the thiazine dye methylene blue asserts its properties as an oxidizing agent only at very high doses, whereas at pharmacologic doses it has reducing agent properties and is for this reason used as a medication for the treatment of methemoglobinemia. A recent laboratory study identified methylene blue as a potent inhibitor of gametocyte development across all stages, almost fully abolishing P. falciparum transmission to mosquitoes at concentrations readily achievable in humans. In addition, a recent clinical study in 180 children with uncomplicated falciparum malaria in Burkina Faso showed that, compared to artesunate-amodiaquine alone, addition of the cheap drug methylene blue to either artesunate or amodiaquine importantly reduced gametocyte carrier rates measured at days 3, 7, and 14 of follow-up. This effect was seen both in patients with and without P. falciparum gametocytaemia at baseline. The current series of studies will investigate further methylene blue as a potential gametocytocidal drug in the treatment of uncomplicated falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

1. For G6PD normal group, healthy males and females as judged by a physician with no abnormality identified on a medical evaluation including medical history and physical examination with laboratory diagnosis of G6PD normal.

   For G6PD deficient group, healthy males with laboratory diagnosis of G6PD deficiency grade 3 with enzyme activity 10-60%.
2. Subjects aged between 18 years to 60 years.
3. Subjects who have Hb ≥ 11 mg/dl.
4. A female is eligible to enter and participate in this study if she is:

   * of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy
   * or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
   * or of childbearing potential, has a negative serum pregnancy test at screening and urine pregnancy test prior to start the study drug in each period, and abstain from sexual intercourse or agrees to using effective contraceptive methods (e.g., intrauterine device, hormonal contraceptive drug, tubal ligation or female barrier method with spermicide) during the study until completion of the follow-up procedures.
5. Read, comprehend, and write at a sufficient level to complete study-related materials.
6. Provide a signed and dated written informed consent prior to study participation.
7. Normal electrocardiogram (ECG) with QTc < 450 msec.
8. Willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. A positive pre-study hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
3. Subjects with a personal history of hypertension, cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de points (heart failure, hypokalemia).
4. Subjects with a family history of sudden cardiac death.
5. A creatinine clearance <70 mL/min as determined by Cockcroft-Gault equation: CLcr (mL/min) = (140 - age) * Wt / (72 * Scr) (multiply answer by 0.85 for females) Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dL [Cockcroft, 1976].
6. History of alcohol or substance abuse or dependence within 6 months of the study: History of regular alcohol consumption averaging >7 drinks/wk for women or >14 drinks/wk for men. One drink is equivalent to 12 g alcohol = 5 oz (150 mL) of wine or 12 oz (360 mL) of beer or 1.5 oz (45 mL) of 80 proof distilled spirits within 6 months of screening.
7. Use of prescription or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety.
8. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
9. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample during each regimen.
10. The subject is unwilling to abstain from the ingestion of grapefruit containing products for 72 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each period.
11. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period. Note: This does not include plasma donation.
12. Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
13. Those who, in the opinion of the investigator, have a risk of non-compliance with study procedures.
14. AST or ALT >1.5 upper limit of normal (ULN).
15. Subjects with history of renal disease, hepatic disease, and/or cholecystectomy.
16. Abnormal methaemoglobin level.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of Primaquine | 7 days
  Maximum concentration (Cmax), Area under the concentration curve (AUC 0-24), Elimination rate constant (PRQ-λz), and Elimination half life (t1/2) for primaquine when given standard dose in G6PD normal and G6PD deficiency
Pharmacokinetic profile of Carboxyprimaquine | 7 days
  Maximum concentration (Cmax), area under the concentration curve (AUC 0-24), elimination rate constant (PRQ-λz), and elimination half life (t1/2) for carboxyprimaquine (primaquine metabolite) when given standard dose in G6PD normal and G6PD deficiency
Pharmacokinetic profile of Methylene blue | 7 days
  Maximum concentration(Cmax), area under the concentration curve (AUC 0-24) elimination rate constant (MB-λz), and elimination half life (t1/2) for methylene blue when given standard dose in G6PD normal and G6PD deficiency
Oocysts production in mosquitoes | 7 days
  Reduction of oocysts production in mosquitoes fed with gametocytes which were exposed to methylene blue and primaquine
Methaemoglobin, Hematocrit and Hemoglobin levels | 7 days
  Methaemoglobin, hematocrit and hemoglobin level when given primaquine and methylene blue in G6PD normal and G6PD deficiency

SECONDARY OUTCOMES:
Safety of Primaquine and Methylene Blue | 1 month
  Safety and tolerability parameters, including adverse events, clinical laboratory, and vital signs assessments

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Tropical Diseases, Bangkok, Thailand